CLINICAL TRIAL: NCT03903848
Title: Immune and Skeletal Muscle Response to an Exercise Session in Cancer Survivors
Brief Title: Cancer Survivors Acute Exercise Response 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Melissa M Markofski, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001419
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms Malignant
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise session (Experimental): One session of physical exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Single session of treadmill walking and resistance exercise

SUMMARY:
The aims of this study examine the immune system, muscle metabolism, and autonomic nervous system response to an acute bout of exercise. Cancer survivors will participate in an acute bout of exercise. Blood samples will be collected before the exercise bout and at two time points after the exercise bout to assess the proposed variables.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-70 years

  * At least two years past detectible cancer (two years disease-free survival)
  * Have received chemotherapy and/or radiation as part of their cancer treatment
  * All cancers were of the organs/non-blood producing tissues (not blood/hematologic cancers) and while they were an adult (no history of pediatric cancer)
  * Meeting ACSM-AHA guidelines for exercise (150 minutes per week of cardiorespiratory fitness type exercises and ~two days per week of resistance training), as confirmed by a combination of a physical activity questionnaire and a cardiorespiratory fitness classification of "good" or higher (age and sex matched)
  * A BMI between 20-33 kg·m-2
  * Able to speak and read English

Exclusion Criteria:

Participants may not:

* Have any contraindications to moderate to vigorous exercise
* Have any recent illness or have been instructed not to exercise by a healthcare provider
* Participants may not have range of motion restrictions that would prevent them from participating in aerobic or resistance training with proper form (they must be ambulatory)
* Be taking medications (prescription or over the counter) known to influence immune function (including daily NSAID's and beta blockers), cholesterol-lowering medications (statins), drugs that increase bone mass (bisphosphonates), or steroids.
* Have known cardiovascular, respiratory, metabolic, or renal disease, with the exception of controlled hypertension (as defined by resting BP below 140/90) and/or controlled asthma (self-reported).
* Be pregnant
* Be unable to complete all visits (i.e. must not be planning to leave the Houston area long-term before concluding their participation in the study)
* Fall outside of a BMI range of (20 - 33)
* Consume alcohol or recreational drugs for 24h prior to visits
* Participants must not have scheduling conflicts that would prevent them from reporting to the laboratory of integrated physiology 2-3 times over the course of the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise-induced response of circulating monocytes | Pre-exercise, change from pre-exercise to immediately post-exercise, change from pre-exercise to 1hr post-exercise, change from immediately post-exercise to 1hr post-exercise
  Circulating serum monocyte phenotype before and after one exercise session
Exercise-induced response of circulating T cells | Pre-exercise, change from pre-exercise to immediately post-exercise, change from pre-exercise to 1hr post-exercise, change from immediately post-exercise to 1hr post-exercise
  Circulating serum T cells phenotype before and after one exercise session
Exercise-induced response of circulating Follistatin | Pre-exercise, change from pre-exercise to immediately post-exercise, change from pre-exercise to 1hr post-exercise, change from immediately post-exercise to 1hr post-exercise
  Circulating serum follistatin before and after one exercise session
Exercise-induced response of circulating GDF-15 | Pre-exercise, change from pre-exercise to immediately post-exercise, change from pre-exercise to 1hr post-exercise, change from immediately post-exercise to 1hr post-exercise
  Circulating serum growth differentiation factor 15 before and after one exercise session

SECONDARY OUTCOMES:
Body composition | before exercise
  Relative body composition, as calculated from a DEXA scan. Measurement will be used as a descriptive variable and potential covariant
Body weight | before exercise
  Absolute body weight as measured with an eye level beam. Measurement will be used as a descriptive variable and potential covariant

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Markofski, Principal Investigator — University of Houston

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared if publication journal requires data sharing
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication
Access Criteria: If when submitting manuscript for publication, the journal requires the release of data then the data will be shared (exact method will be consistent with journal policy, but may include inclusion as a supplementary figure or depositing in a data repository suggested by the journal)